CLINICAL TRIAL: NCT02832336
Title: The Effect of Caffeine on the Narcoleptic Patients Randomized Controlled Clinical Trial
Brief Title: The Effect of Caffeine on the Narcoleptic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: King Saud Medical City (Other Government)
Responsible Party: Principal Investigator, Mona Aldoasri, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB:E-15-1484; SFDA # 16022302 (Registry Identifier: Saudi Clinical Trials Registry)
Record Dates: First submitted 2016-06-09; First posted 2016-07-14 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Narcolepsy
Keywords: Caffeine; Caffeine citrate; Neurological disorder; Excessive daytime sleepiness; Orexin; adenosine antagonist
MeSH Terms: conditions — Narcolepsy; Nervous System Diseases; Disorders of Excessive Somnolence | interventions — Caffeine; caffeine citrate; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caffeine (Experimental): Caffeine is an adenosine receptor antagonist. It inhibits a part of the sleep cycle and, in turn, promotes the wakefulness state.
  Generic name :Vivarin(1,3,7-trimethylxanthine), 200 mg/day for one week, Form of Administration:Oral in veg white capsule form (size 1) Drug Class:Central nervous system (CNS) stimulants.
  Interventions: Drug: Vivarin
- Fiber (Placebo Comparator): Fiber powder will be used as placebo, Form of Administration:Oral in veg white capsule form (size 1)
  Interventions: Drug: Fiber

INTERVENTIONS:
Drug: Vivarin — Adenosine is an endogenous sleep-promoting substance with neuronal inhibitory effects. Adenosine has been proposed to be a sleep-inducing substance accumulating in the brain during prolonged wakefulness. Caffeine is an adenosine receptor antagonist. It inhibits a part of the sleep cycle and, in turn, promotes the wakeup state. Caffeine results in the release of norepinephrine, dopamine and serotonin in the brain and the increase of circulating catecholamines, consistent with reversal of the inhibitory effect of adenosine.Vivarin Drug class :Central nervous system (CNS) stimulants.
  Other Names: 1,3,7-Trimethylpurine-2,6-dione; C8H10N4O2; caffeine citrate
  Arms: Caffeine
Drug: Fiber — Fiber will be used as placebo.
  Other Names: Nutrisource Fiber
  Arms: Fiber

SUMMARY:
Caffeine may be playing a beneficial role in patients with narcolepsy. However, the relationship between caffeine and its effects on narcoleptic patients has not been examined, and it is also unclear whether caffeine provides a beneficial effect or not. Hence, the aim of this study is to assess the effects of caffeine consumption on daytime sleepiness and reaction time in narcoleptic patients.

DETAILED DESCRIPTION:
The participants will be recruited at the University Sleep Disorders Center, College of Medicine, King Saud University.

Narcolepsy diagnosis: Narcolepsy will be diagnosed based on the American Academy of Sleep Medicine International Classification of Sleep Disorders, 2014 (American academy of sleep medicine. International classification of sleep disorders (ICSD), 3rd ed. Darien, il: American academy of sleep medicine, 2014).

The study will be interventional, randomized, double-blind, placebo control study, to evaluate the effect of caffeine on Narcoleptic Adults (n=30) aged 18-45 years old, following up in the Sleep Disorders Center (SDC) at King Khalid University Hospital (KKUH).

Tools of the study:

The study tools included an interview questionnaire, anthropometric measurements, indirect calorimetry, body composition measurements, blood biochemistry tests & Eye Blink measurement.

1. Interview Questionnaire:

   For collecting data for this study, questionnaire well be designed.

   The questionnaire consisted of four parts to elicit the following information:

   A) Socio-demographic Data
   * Personal data: The name of the participant, age, sex, educational level, and residence.
   * Social habits: The smoking status
   * Activity level: Mild, moderate or intense physical activity.

   B) Medical information:
   * The occurrence of Narcolepsy with or without cataplexy.
   * The occurrence of chronic diseases (hypertension, hyperlipidemia, cardiac diseases, diabetes and obesity).

   C) Caffeine expectancy & consumption, modified from:
   * Caffeine expectancy questionnaire (CaffEQ) is a self-report measure, which assesses a range of expectancies for caffeine, and Sleep Disturbance (Huntley & Juliano, 2007).
   * The Caffeine Consumption Questionnaire (CCQ) used to produce a typical week's average estimate of caffeine consumption in milligrams (Heaton, 2010).

   D) Daytime sleepiness Scales :
   * Stanford Sleepiness Scale (SSS)
   * The Karolinska Sleepiness Scale (KSS)
2. Anthropometric measurements:

   The four selected anthropometric measures, see below:
   * Weight
   * Height for calculating body mass index (BMI)
   * Waist circumference
   * Hip circumference
3. Indirect calorimetry An automated metabolic measuring cart used for determining Energy Expenditure and for providing key information about the nutrient mixture catabolized for energy by measuring the rates of O2 consumption (VO2) and CO2 production (VCO2), the device name is QUARK.
4. Body Composition Measurement:

   The five variables selected for body composition measurements are:
   * Fat mass
   * Muscle mass
   * Bone mass
   * Total body water
   * Visceral fat rating The body composition machine will be used is Bioelectrical impedance analysis (Tanita BC-418, Japan).
5. Blood biochemistry tests:

   Fasting blood glucose, lipids Profile, CBC, LFT, CRP, Bone Profile, Vit D. Biochemical measurements will be done at KKUH, it is equipped with all needed matching to run this study and has well-trained technician and statics to help in performing the test needed.
6. Eye Blink Measurement. Setting/Procedure

In the day of study, subject need to come fasting overnight so their fasting blood glucose levels and lab test sample will be taken. Then the Anthropometric, Body Composition & Indirect calorimetry Measurement for the subject will be documented. The sample will be randomly divided using a software and the tablets will be identically packaged by the pharmacist in opaque capsules and administered orally in a double- blind setting to one of the following Groups:

* Group one: will receive 200 mg Caffeine capsule + water.
* Group two: will receive Placebo (fiber capsule) + water.

Then instruct the patients to take the medication/placebo in the morning for 1 week and come back for reassessment:

* Random Blood sugar will be taken
* Blood Pressure will be measured.
* Eye Blink Measurement
* Daytime sleepiness Scales (part of the questioner data will be filled) We will have a baseline assessment, 1st assessment after single dose of 200 mg Caffeine or placebo and second assessment after one week of chronic use of medication in a dose 200 mg During the patient waiting time, the Interview Questionnaire will be filled.

Data management:

Data will be categorized to age, sex, social, anthropometric measurements, biochemistry lab test, psychological and medical status.

Statistical analysis Data will be entered and statistically analyzed by SPSS software. ANOVA will be used to differentiate among treatment groups. In all the statistical comparisons, differences with p < 0.05 will be considered to be significant.

Steps for assuring data quality include:

* Training: Educate data collectors in a structured manner.
* Data completeness: Using the hospital program (Cerner) that give immediate feedback on issues such as missing or out-of-range values & Excel software
* Data consistency: Compare across sites and over time.
* Data dictionary will be used e.g World Health Organization Drug Dictionary, Cerner program record for normal ranges.

Ethical consideration The study was approved by KKUH Ethical committee, Saudi Food & Drug Authority & Saudi Clinical Trial Registry.

ELIGIBILITY:
Inclusion Criteria:

* Case -group should be Narcoleptic with cataplexy

Exclusion Criteria:

* Individuals older than 45 years or younger than 18 years old.
* Individuals complaining of any diseases or conditions that affect their dietary intake, as such : renal failure, liver failure, malabsorption problems, cardiac diseases … etc.
* Individuals having hypersensitivity to caffeine.
* Individuals with medical conditions that cause sleepiness (like hypothyroidism) and pregnant or lactating females will be excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-10-01; Primary Completion 2017-05-11 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Eye Blink Measurement | 7 days
  Blink total duration (BTD), which measures the duration of the closing, closed and reopening phases of each blink by using Optalert system, a glass frame carrying an IR transmitter and receiver bar that positioned below and in front of the eye, directed towards the lower edge of the upper eyelid allows for measurements of blink duration and eye closure time as an indicator of drowsiness and decreased vigilance.The eye blink measurement (Optalert) will be performed multiple times to measure the changes in the alertness level for each patient after single-dose intake and after daily medication intake.(The measuring instrument takes about 10-20 minutes).

SECONDARY OUTCOMES:
Stanford Sleepiness Scale (SSS) | 7 days
  SSS is a daytime sleepiness Scales, using a 7-point Likert scale based on a series of statements that range from "feeling active, vital, alert, wide awake" to "almost in reverie, cannot stay awake, sleep onset appears imminent" describes how they feel at the time (Hoddes et.al,1973).
The Karolinska Sleepiness Scale (KSS) | 7 days
  KSS is a daytime sleepiness Scales, using a 9-point Likert scale based on a self-reported, subjective assessment of the subject's level of drowsiness at the time (Akerstedt & Gillberg, 1990).

CONTACTS AND LOCATIONS:
Overall Officials: Mona S Aldosari, Masteral, Principal Investigator — King Saud University
Locations (1):
- King Khalid University Hospital:King Saud Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
Possibility to share most data.

REFERENCES:
- [Background] Adamantidis AR, Zhang F, Aravanis AM, Deisseroth K, de Lecea L. Neural substrates of awakening probed with optogenetic control of hypocretin neurons. Nature. 2007 Nov 15;450(7168):420-4. doi: 10.1038/nature06310. Epub 2007 Oct 17. PMID 17943086
- [Background] Akerstedt T, Gillberg M. Subjective and objective sleepiness in the active individual. Int J Neurosci. 1990 May;52(1-2):29-37. doi: 10.3109/00207459008994241. PMID 2265922
- [Background] Alkaabi J, Al-Dabbagh B, Saadi H, Gariballa S, Yasin J. Effect of traditional Arabic coffee consumption on the glycemic index of Khalas dates tested in healthy and diabetic subjects. Asia Pac J Clin Nutr. 2013;22(4):565-73. doi: 10.6133/apjcn.2013.22.4.09. PMID 24231017
- [Background] BaHammam AS, Alenezi AM. Narcolepsy in Saudi Arabia. Demographic and clinical perspective of an under-recognized disorder. Saudi Med J. 2006 Sep;27(9):1352-7. PMID 16951772
- [Background] Beitinger PA, Fulda S, Dalal MA, Wehrle R, Keckeis M, Wetter TC, Han F, Pollmacher T, Schuld A. Glucose tolerance in patients with narcolepsy. Sleep. 2012 Feb 1;35(2):231-6. doi: 10.5665/sleep.1628. PMID 22294813
- [Background] Benowitz NL. Clinical pharmacology of caffeine. Annu Rev Med. 1990;41:277-88. doi: 10.1146/annurev.me.41.020190.001425. PMID 2184730
- [Background] Bruck D, Armstrong S, Coleman G. Sleepiness after glucose in narcolepsy. J Sleep Res. 1994 Sep;3(3):171-179. doi: 10.1111/j.1365-2869.1994.tb00125.x. PMID 10607123
- [Background] Burdakov D, Alexopoulos H. Metabolic state signalling through central hypocretin/orexin neurons. J Cell Mol Med. 2005 Oct-Dec;9(4):795-803. doi: 10.1111/j.1582-4934.2005.tb00380.x. PMID 16364191
- [Background] Chabas D, Foulon C, Gonzalez J, Nasr M, Lyon-Caen O, Willer JC, Derenne JP, Arnulf I. Eating disorder and metabolism in narcoleptic patients. Sleep. 2007 Oct;30(10):1267-73. doi: 10.1093/sleep/30.10.1267. PMID 17969460
- [Background] Chemelli RM, Willie JT, Sinton CM, Elmquist JK, Scammell T, Lee C, Richardson JA, Williams SC, Xiong Y, Kisanuki Y, Fitch TE, Nakazato M, Hammer RE, Saper CB, Yanagisawa M. Narcolepsy in orexin knockout mice: molecular genetics of sleep regulation. Cell. 1999 Aug 20;98(4):437-51. doi: 10.1016/s0092-8674(00)81973-x. PMID 10481909
- [Background] Cun Y, Tang L, Yan J, He C, Li Y, Hu Z, Xia J. Orexin A attenuates the sleep-promoting effect of adenosine in the lateral hypothalamus of rats. Neurosci Bull. 2014 Oct;30(5):877-86. doi: 10.1007/s12264-013-1442-8. Epub 2014 Jun 5. PMID 24898402
- [Background] Dahmen N, Bierbrauer J, Kasten M. Increased prevalence of obesity in narcoleptic patients and relatives. Eur Arch Psychiatry Clin Neurosci. 2001;251(2):85-9. doi: 10.1007/s004060170057. PMID 11407443
- [Background] Daniels E, King MA, Smith IE, Shneerson JM. Health-related quality of life in narcolepsy. J Sleep Res. 2001 Mar;10(1):75-81. doi: 10.1046/j.1365-2869.2001.00234.x. PMID 11285058
- [Background] Daniello A, Fievisohn E, Gregory TS. Modeling the effects of caffeine on the sleep/ wake cycle. Biomed Sci Instrum. 2012;48:73-80. PMID 22846267
- [Background] Darwish M, Kirby M, Robertson P Jr, Hellriegel ET. Interaction profile of armodafinil with medications metabolized by cytochrome P450 enzymes 1A2, 3A4 and 2C19 in healthy subjects. Clin Pharmacokinet. 2008;47(1):61-74. doi: 10.2165/00003088-200847010-00006. PMID 18076219
- [Background] Dresler M, Spoormaker VI, Beitinger P, Czisch M, Kimura M, Steiger A, Holsboer F. Neuroscience-driven discovery and development of sleep therapeutics. Pharmacol Ther. 2014 Mar;141(3):300-34. doi: 10.1016/j.pharmthera.2013.10.012. Epub 2013 Nov 1. PMID 24189488
- [Background] Engel A, Helfrich J, Manderscheid N, Musholt PB, Forst T, Pfutzner A, Dahmen N. Investigation of insulin resistance in narcoleptic patients: dependent or independent of body mass index? Neuropsychiatr Dis Treat. 2011;7:351-6. doi: 10.2147/NDT.S18455. Epub 2011 Jun 9. PMID 21822386
- [Background] Espana RA, McCormack SL, Mochizuki T, Scammell TE. Running promotes wakefulness and increases cataplexy in orexin knockout mice. Sleep. 2007 Nov;30(11):1417-25. doi: 10.1093/sleep/30.11.1417. PMID 18041476
- [Background] Flygare J, Parthasarathy S. Narcolepsy: let the patient's voice awaken us! Am J Med. 2015 Jan;128(1):10-3. doi: 10.1016/j.amjmed.2014.05.037. Epub 2014 Jun 12. PMID 24931392
- [Background] Hoddes E, Zarcone V, Smythe H, Phillips R, Dement WC. Quantification of sleepiness: a new approach. Psychophysiology. 1973 Jul;10(4):431-6. doi: 10.1111/j.1469-8986.1973.tb00801.x. No abstract available. PMID 4719486
- [Background] Honda Y, Doi Y, Ninomiya R, Ninomiya C. Increased frequency of non-insulin-dependent diabetes mellitus among narcoleptic patients. Sleep. 1986;9(1 Pt 2):254-9. doi: 10.1093/sleep/9.1.254. PMID 3518018
- [Background] Ingravallo F, Gnucci V, Pizza F, Vignatelli L, Govi A, Dormi A, Pelotti S, Cicognani A, Dauvilliers Y, Plazzi G. The burden of narcolepsy with cataplexy: how disease history and clinical features influence socio-economic outcomes. Sleep Med. 2012 Dec;13(10):1293-300. doi: 10.1016/j.sleep.2012.08.002. Epub 2012 Sep 28. PMID 23026503
- [Background] Jennum P, Ibsen R, Knudsen S, Kjellberg J. Comorbidity and mortality of narcolepsy: a controlled retro- and prospective national study. Sleep. 2013 Jun 1;36(6):835-40. doi: 10.5665/sleep.2706. PMID 23729926
- [Background] Johnston KL, Clifford MN, Morgan LM. Coffee acutely modifies gastrointestinal hormone secretion and glucose tolerance in humans: glycemic effects of chlorogenic acid and caffeine. Am J Clin Nutr. 2003 Oct;78(4):728-33. doi: 10.1093/ajcn/78.4.728. PMID 14522730
- [Background] Kaplan GB, Greenblatt DJ, Ehrenberg BL, Goddard JE, Cotreau MM, Harmatz JS, Shader RI. Dose-dependent pharmacokinetics and psychomotor effects of caffeine in humans. J Clin Pharmacol. 1997 Aug;37(8):693-703. doi: 10.1002/j.1552-4604.1997.tb04356.x. PMID 9378841
- [Background] Landolt HP. Sleep homeostasis: a role for adenosine in humans? Biochem Pharmacol. 2008 Jun 1;75(11):2070-9. doi: 10.1016/j.bcp.2008.02.024. Epub 2008 Mar 4. PMID 18384754
- [Background] Landolt HP, Retey JV, Tonz K, Gottselig JM, Khatami R, Buckelmuller I, Achermann P. Caffeine attenuates waking and sleep electroencephalographic markers of sleep homeostasis in humans. Neuropsychopharmacology. 2004 Oct;29(10):1933-9. doi: 10.1038/sj.npp.1300526. PMID 15257305
- [Background] Longstreth WT Jr, Koepsell TD, Ton TG, Hendrickson AF, van Belle G. The epidemiology of narcolepsy. Sleep. 2007 Jan;30(1):13-26. doi: 10.1093/sleep/30.1.13. PMID 17310860
- [Background] Mesa YR, Meira E Cruz MG. Narcolepsy with cataplexy after A/H1N1 vaccination - A case reported from Cuba. Sleep Sci. 2014 Mar;7(1):59-61. doi: 10.1016/j.slsci.2014.07.024. Epub 2014 Aug 22. PMID 26483903
- [Background] Nawrot P, Jordan S, Eastwood J, Rotstein J, Hugenholtz A, Feeley M. Effects of caffeine on human health. Food Addit Contam. 2003 Jan;20(1):1-30. doi: 10.1080/0265203021000007840. PMID 12519715
- [Background] Partinen M, Saarenpaa-Heikkila O, Ilveskoski I, Hublin C, Linna M, Olsen P, Nokelainen P, Alen R, Wallden T, Espo M, Rusanen H, Olme J, Satila H, Arikka H, Kaipainen P, Julkunen I, Kirjavainen T. Increased incidence and clinical picture of childhood narcolepsy following the 2009 H1N1 pandemic vaccination campaign in Finland. PLoS One. 2012;7(3):e33723. doi: 10.1371/journal.pone.0033723. Epub 2012 Mar 28. PMID 22470463
- [Background] Peacock J, Benca RM. Narcolepsy: clinical features, co-morbidities & treatment. Indian J Med Res. 2010 Feb;131:338-49. PMID 20308759
- [Background] Peall KJ, Robertson NP. Narcolepsy: environment, genes and treatment. J Neurol. 2014 Aug;261(8):1644-6. doi: 10.1007/s00415-014-7435-3. No abstract available. PMID 25034273
- [Background] Plaza-Zabala A, Maldonado R, Berrendero F. The hypocretin/orexin system: implications for drug reward and relapse. Mol Neurobiol. 2012 Jun;45(3):424-39. doi: 10.1007/s12035-012-8255-z. Epub 2012 Mar 20. PMID 22430644
- [Background] Poli F, Plazzi G, Di Dalmazi G, Ribichini D, Vicennati V, Pizza F, Mignot E, Montagna P, Pasquali R, Pagotto U. Body mass index-independent metabolic alterations in narcolepsy with cataplexy. Sleep. 2009 Nov;32(11):1491-7. doi: 10.1093/sleep/32.11.1491. PMID 19928388
- [Background] al Rajeh S, Bademosi O, Ismail H, Awada A, Dawodu A, al-Freihi H, Assuhaimi S, Borollosi M, al-Shammasi S. A community survey of neurological disorders in Saudi Arabia: the Thugbah study. Neuroepidemiology. 1993;12(3):164-78. doi: 10.1159/000110316. PMID 8272177
- [Background] Sakurai T, Amemiya A, Ishii M, Matsuzaki I, Chemelli RM, Tanaka H, Williams SC, Richardson JA, Kozlowski GP, Wilson S, Arch JR, Buckingham RE, Haynes AC, Carr SA, Annan RS, McNulty DE, Liu WS, Terrett JA, Elshourbagy NA, Bergsma DJ, Yanagisawa M. Orexins and orexin receptors: a family of hypothalamic neuropeptides and G protein-coupled receptors that regulate feeding behavior. Cell. 1998 Feb 20;92(4):573-85. doi: 10.1016/s0092-8674(00)80949-6. PMID 9491897
- [Background] Sakurai T, Mieda M, Tsujino N. The orexin system: roles in sleep/wake regulation. Ann N Y Acad Sci. 2010 Jul;1200:149-61. doi: 10.1111/j.1749-6632.2010.05513.x. PMID 20633143
- [Background] Sasaki K, Suzuki M, Mieda M, Tsujino N, Roth B, Sakurai T. Pharmacogenetic modulation of orexin neurons alters sleep/wakefulness states in mice. PLoS One. 2011;6(5):e20360. doi: 10.1371/journal.pone.0020360. Epub 2011 May 27. PMID 21647372
- [Background] Sellayah D, Bharaj P, Sikder D. Orexin is required for brown adipose tissue development, differentiation, and function. Cell Metab. 2011 Oct 5;14(4):478-90. doi: 10.1016/j.cmet.2011.08.010. PMID 21982708
- [Background] Serra L, Montagna P, Mignot E, Lugaresi E, Plazzi G. Cataplexy features in childhood narcolepsy. Mov Disord. 2008 Apr 30;23(6):858-65. doi: 10.1002/mds.21965. PMID 18307264
- [Background] Sicard BA, Perault MC, Enslen M, Chauffard F, Vandel B, Tachon P. The effects of 600 mg of slow release caffeine on mood and alertness. Aviat Space Environ Med. 1996 Sep;67(9):859-62. PMID 9025802
- [Background] Silber MH, Krahn LE, Olson EJ, Pankratz VS. The epidemiology of narcolepsy in Olmsted County, Minnesota: a population-based study. Sleep. 2002 Mar 15;25(2):197-202. doi: 10.1093/sleep/25.2.197. PMID 11902429
- [Background] Thorpy MJ, Krieger AC. Delayed diagnosis of narcolepsy: characterization and impact. Sleep Med. 2014 May;15(5):502-7. doi: 10.1016/j.sleep.2014.01.015. Epub 2014 Feb 15. PMID 24780133
- [Background] Wesensten NJ, Belenky G, Thorne DR, Kautz MA, Balkin TJ. Modafinil vs. caffeine: effects on fatigue during sleep deprivation. Aviat Space Environ Med. 2004 Jun;75(6):520-5. PMID 15198278
- [Background] Wright KP Jr, Badia P, Myers BL, Plenzler SC. Combination of bright light and caffeine as a countermeasure for impaired alertness and performance during extended sleep deprivation. J Sleep Res. 1997 Mar;6(1):26-35. doi: 10.1046/j.1365-2869.1997.00022.x. PMID 9125696
- [Background] Won C, Mahmoudi M, Qin L, Purvis T, Mathur A, Mohsenin V. The impact of gender on timeliness of narcolepsy diagnosis. J Clin Sleep Med. 2014 Jan 15;10(1):89-95. doi: 10.5664/jcsm.3370. PMID 24426826
- [Background] Zhang N, Liu HT. Effects of sleep deprivation on cognitive functions. Neurosci Bull. 2008 Feb;24(1):45-8. doi: 10.1007/s12264-008-0910-z. PMID 18273076
- [Background] Zhang XY, Yu L, Zhuang QX, Zhu JN, Wang JJ. Central functions of the orexinergic system. Neurosci Bull. 2013 Jun;29(3):355-65. doi: 10.1007/s12264-012-1297-4. Epub 2013 Jan 8. PMID 23299718
- [Derived] Aldosari MS, Olaish AH, Nashwan SZ, Abulmeaty MMA, BaHammam AS. The effects of caffeine on drowsiness in patients with narcolepsy: a double-blind randomized controlled pilot study. Sleep Breath. 2020 Dec;24(4):1675-1684. doi: 10.1007/s11325-020-02065-6. Epub 2020 Mar 26. PMID 32215834